CLINICAL TRIAL: NCT07114835
Title: Investigation of the Effects of Low-Intensity Cycling Exercise Combined With Blood Flow Restriction on VO2max, Muscle Strength, and Muscle Thickness in Physically Active Individuals
Brief Title: Low-Intensity BFR Cycling: Impact on VO₂Max and Muscle Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Gönül YAVUZ, Asisst. Prof., Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BFR-Cycling-2025
Record Dates: First submitted 2025-06-30; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Aerobic Capacity; Blood Flow Restriction (BFR) Training Effects; Blood Flow Restriction Exercise; Muscle Strengh; Isokinetic; VO2max
Keywords: Blood flow restriction; aerobic capacity; VO2max; muscle strength; muscle thickness

STUDY DESIGN:
Intervention Model Description: Initially, 30 male volunteers who were not actively engaged in sports were recruited for the study. After applying the exclusion criteria, which included a history of lower extremity injury (n = 4), respiratory disorders (n = 1) and refusal to participate (n = 1), a total of six individuals were excluded in the initial phase. Thus, the study commenced with 24 male participants. Each group consisted of eight participants who completed the protocol and final post-tests were conducted and analysed accordingly. All participants were healthy individuals who did not engage in regular physical activity. The study involved three exercise groups: The Control Group (CG); the Cycling with Blood Flow Restriction Group (CBFRG); Cycling Exercise Group (CEG)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cycling Exercise - 40 min at 40% VO₂max (Experimental): Participants in this group perform low-intensity cycling exercise at 40% of their VO₂max for 40 minutes per session, three times per week, over a 9-week period. All sessions are conducted on an electronically braked Astrand cycle ergometer. This group does not receive blood flow restriction.
  Interventions: Procedure: Cycling Exercise (40 min at 40% VO₂max)
- Control - 15 min Cycling at 40% VO₂max (Active Comparator): Participants in the control group perform cycling exercise at 40% of their VO₂max for 15 minutes per session, three times per week for 9 weeks. The exercise is performed on an electronically braked Astrand cycle ergometer. No blood flow restriction or additional intervention is applied in this group.
  Interventions: Procedure: Short-Duration Cycling Control (15 min at 40% VO₂max)
- Cycling + BFR - 15 min at 40% VO₂max with 60-80% LOP (Experimental): Participants in this group perform cycling exercise at 40% of their VO₂max for 15 minutes per session, three times per week for 9 weeks. During each session, pneumatic cuffs are applied to the proximal thighs to restrict blood flow, with individualized limb occlusion pressure (LOP) set at 60% in weeks 1-4, 70% in weeks 5-7, and 80% in weeks 8-9. The exercise is performed on an electronically braked Astrand cycle ergometer.
  Interventions: Procedure: Cycling with Blood Flow Restriction (15 min at 40% VO₂max with 60-80% LOP)

INTERVENTIONS:
Procedure: Cycling with Blood Flow Restriction (15 min at 40% VO₂max with 60-80% LOP) — This intervention involves low-intensity cycling exercise at 40% of VO₂max performed on an electronically braked Astrand cycle ergometer for 15 minutes per session. During each session, pneumatic cuffs (10 cm wide, manually adjustable) are applied to the upper thighs to restrict blood flow. Individualized limb occlusion pressure (LOP) is determined via Doppler ultrasound and set progressively at 60% (weeks 1-4), 70% (weeks 5-7), and 80% (weeks 8-9). Sessions are conducted three times per week over a 9-week period. The aim is to simulate the physiological effects of high-intensity training using a low-intensity protocol.
  Other Names: BFR Cycling; Low-Intensity Cycling + BFR; CBFR
  Arms: Cycling + BFR - 15 min at 40% VO₂max with 60-80% LOP
Procedure: Cycling Exercise (40 min at 40% VO₂max) — This intervention involves standard low-intensity cycling exercise at 40% of the participant's VO₂max, performed for 40 minutes per session on an electronically braked Astrand cycle ergometer. Sessions are conducted three times per week for a total duration of 9 weeks. This group does not receive any blood flow restriction or external loading. The aim is to observe the effects of traditional low-intensity, long-duration aerobic exercise on VO₂max, muscle strength, and muscle thickness.
  Other Names: CEG; Standard Low-Intensity Cycling; Long-duration Cycling
  Arms: Cycling Exercise - 40 min at 40% VO₂max
Procedure: Short-Duration Cycling Control (15 min at 40% VO₂max) — This intervention involves low-intensity cycling exercise at 40% of VO₂max performed for 15 minutes per session, using an electronically braked Astrand cycle ergometer. Participants exercise three times per week for 9 weeks. No blood flow restriction is applied. The aim of this control condition is to match the duration of the BFR intervention while omitting the occlusion component, to isolate the effect of BFR.
  Other Names: Control Group Cycling; CG Short Cycling; No BFR
  Arms: Control - 15 min Cycling at 40% VO₂max

SUMMARY:
This study aims to investigate the effects of low-intensity cycling exercise combined with blood flow restriction (BFR) on maximal oxygen consumption (VO₂max), muscle strength, and muscle thickness in sedentary adult males. Participants will be randomly assigned to three groups: (1) a cycling exercise group performing 40 minutes of cycling at 40% VO₂max, (2) a cycling with blood flow restriction group performing 15 minutes of cycling at 40% VO₂max with limb occlusion pressure at 60-80%, and (3) a control group following a shorter cycling protocol. Muscle thickness, isokinetic knee strength, and VO₂max will be measured before and after the 9-week intervention. The study is designed to evaluate whether short-duration, low-intensity cycling with BFR can induce physiological adaptations comparable to traditional longer-duration cycling protocols.

DETAILED DESCRIPTION:
This study is designed to examine the effects of low-intensity cycling exercise combined with blood flow restriction (BFR) on aerobic capacity (VO₂max), isokinetic knee strength, and muscle thickness in sedentary male adults. Traditional methods for improving aerobic capacity and muscle strength often involve high-intensity or long-duration training protocols. However, such protocols may not be feasible for all individuals, particularly during rehabilitation, periods of detraining, or in populations with limited exercise tolerance.

Blood flow restriction training has gained attention as a promising strategy to elicit muscular and cardiovascular adaptations using lower intensities. The technique involves applying individualized limb occlusion pressure (LOP) via pneumatic cuffs during exercise to partially restrict arterial inflow and fully restrict venous outflow. This restriction is thought to create a hypoxic environment and increase metabolic stress, which may enhance the recruitment of fast-twitch muscle fibers and stimulate physiological adaptations.

In this randomized controlled trial, participants are allocated to one of three groups: a standard cycling exercise group (40 minutes at 40% VO₂max), a BFR cycling group (15 minutes at 40% VO₂max with 60-80% LOP), and a control group (15 minutes at 40% VO₂max without BFR). All exercise sessions are performed three times per week for nine weeks. The LOP is adjusted across the training period to progressively increase the stimulus in the BFR group.

Baseline and post-intervention assessments include measurements of body height and weight, ultrasound-based muscle thickness, isokinetic knee strength testing, and graded exercise testing for VO₂max. The goal is to determine whether low-intensity, short-duration cycling with BFR can serve as a practical and effective alternative to longer-duration exercise programs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18-24 years,
* Individuals without any health problems,
* Individuals who do not actively participate in sports,
* Individuals who marked all items as no on the H+cuff participant information form,
* Individuals who have not had a sports injury that would prevent them from participating in sports in the last 6 months,

Exclusion Criteria:

* history of lower extremity injury, respiratory disorders and refusal to participate

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Change in Maximal Oxygen Consumption (VO₂max, L/min) | Baseline and Post-test (Week 9)
  Absolute VO₂max will be measured during a graded cycling exercise test using a breath-by-breath gas analyzer.
Change in Relative VO₂max (ml/kg/min) | Baseline and Post-test (Week 9)
  VO₂max will also be reported relative to body weight using standard calculation: (VO₂max ÷ body weight).

SECONDARY OUTCOMES:
Change in Muscle Thickness (Rectus Femoris, Vastus Lateralis, Biceps Femoris) | Baseline and Post-test (Week 9)
  Muscle thickness will be measured using B-mode ultrasonography with linear probe at specified anatomical landmarks.
Change in Peak Torque (Isokinetic Knee Strength, 60°/s and 180°/s) | Baseline and Post-test (Week 9)
  Isokinetic knee extension and flexion strength will be measured using an isokinetic dynamometer at angular velocities of 60°/s and 180°/s.
Change in Respiratory Exchange Ratio (RER) | Baseline and Post-test (Week 9)
  RER will be recorded during the maximal exercise test as the ratio of carbon dioxide output to oxygen uptake (VCO₂/VO₂).
Change in Maximal Heart Rate (MHR) | Baseline and Post-test (Week 9)
  Maximal heart rate will be recorded during the graded exercise test.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sport Science, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share the results of the training so that they can see their own development and the increase in their performance.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Bennett H, Slattery F. Effects of Blood Flow Restriction Training on Aerobic Capacity and Performance: A Systematic Review. J Strength Cond Res. 2019 Feb;33(2):572-583. doi: 10.1519/JSC.0000000000002963. PMID 30531417
- [Background] Gao Z, Li Y, Zhang J, Li L, Wang T, Wang X, Wang H. Effects of aerobic training with blood flow restriction on aerobic capacity, muscle strength, and hypertrophy in young adults: a systematic review and meta-analysis. Front Physiol. 2025 Jan 7;15:1506386. doi: 10.3389/fphys.2024.1506386. eCollection 2024. PMID 39839525
- [Background] Zeng Q, Wang L, Zhang Y, Wei H, He Z. Effects of blood flow restriction cycling training on body composition and blood lipids in overweight male college students. Front Physiol. 2022;12:792756. doi:10.3389/fphys.2021.792756 22.
- [Result] Abe T, Kearns CF, Sato Y. Muscle size and strength are increased following walk training with restricted venous blood flow from the leg muscle, Kaatsu-walk training. J Appl Physiol (1985). 2006 May;100(5):1460-6. doi: 10.1152/japplphysiol.01267.2005. Epub 2005 Dec 8. PMID 16339340
- [Result] Abe T, Fujita S, Nakajima T, Sakamaki M, Ozaki H, Ogasawara R, Sugaya M, Kudo M, Kurano M, Yasuda T, Sato Y, Ohshima H, Mukai C, Ishii N. Effects of Low-Intensity Cycle Training with Restricted Leg Blood Flow on Thigh Muscle Volume and VO2MAX in Young Men. J Sports Sci Med. 2010 Sep 1;9(3):452-8. eCollection 2010. PMID 24149640

DOCUMENTS (2):
  • Informed Consent Form: Ethics Committee (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT07114835/ICF_000.pdf
  • Informed Consent Form: Ethics Committee Turkish (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT07114835/ICF_001.pdf